CLINICAL TRIAL: NCT02466997
Title: Efficacy of Tacrolimus Ointment 0.1% Versus Placebo in Adults With Facial Non-segmental Vitiligo: a Randomized Double-blind Controlled Study
Brief Title: Efficacy of Tacrolimus in Adults With Facial Non-segmental Vitiligo - VITAC
Acronym: VITAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUBX 2012/05
Record Dates: First submitted 2015-05-26; First posted 2015-06-09 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Vitiligo
Keywords: Vitiligo; Tacrolimus; Face
MeSH Terms: conditions — Vitiligo; Facies | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus group (Experimental): Target-lesion will be treated with the study treatment BID. The batch of treatment (Tacrolimus ointment 0.1% or placebo) will be randomized. All the patients will be treated during 6 months. Counselling on natural daylight exposition will also be given to all patients. During the 6-month observation period, relapse (worsening of VASI ≥ 25%) will be re-treated by the study treatment
  Interventions: Drug: tacrolimus
- Control group (Placebo Comparator): In the Control group, patients will receive the placebo ointment to be applied twice a day during 24 weeks.
  Counselling on natural light exposure during the duration of the trial will be given.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tacrolimus — tacrolimus 0.1% ointment applied twice a day for the experimental group during 24 weeks placebo ointment applied twice a day for the control group during 24 weeks
  Other Names: Protopic
  Arms: Tacrolimus group
Drug: Placebo
  Arms: Control group

SUMMARY:
Multicentric French parallel double-blind randomized versus placebo study

DETAILED DESCRIPTION:
Multicentric French parallel double-blind randomized versus placebo study, with duration of treatment of 6 months, and a post-treatment follow-up period of 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Subject male or female with age over 18 years old
2. Diagnosis of non-segmental (symmetrical) vitiligo
3. Presence of at least one vitiligo target-plaque on the face, with:

   Area greater than 3cm² Local Vitiligo Area Severity Index (VASI) score ≥ 50% Stable (no change in pigmentation or size over the last 3 months) Recent onset (less than 2 years duration)
4. Subject affiliated to the French social security system

Exclusion Criteria:

1. Progressive vitiligo over the last 3 months
2. Spontaneous ongoing repigmentation (documented in the last 3 months)
3. Previous topical Tacrolimus treatment in the last 3 months
4. Previous topical or systemic treatment in the last month:

   Topical or oral corticosteroid Topical vitamin D Phototherapy or laser Other topical treatment specific to vitiligo Other immunosuppressant or immunomodulator
5. Underlying dermatological disease (i.e.: history of atopic dermatitis, eczema, psoriasis), which, according to the investigator, could interfere with the study assessments
6. Known sensitivity to study drug or macrolides
7. Past history of skin cancer or lymphoma
8. Congenital or acquired immunodeficiency
9. Pregnant or breastfeeding women
10. Women without contraception
11. Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of repigmented surface area of the target lesion ≥75% | One year
  To test the efficacy of a 24 weeks months Tacrolimus 0.1% ointment treatment vs placebo in an adult population with stable non-segmental vitiligo of the face. Therapeutic success is defined as the variation in percentage of repigmented surface area of the target lesion ≥75% at 24 weeks months.

SECONDARY OUTCOMES:
Variation in percentage of repigmented surface area | 24 weeks
  Variation in percentage of repigmented surface area of the target lesion between week 24 and week 48 (observation period) in patients who were successfully treated (observation period)
Variation in percentage of repigmented surface area | 48 weeks
  Variation in percentage of repigmented surface area of the target lesion between week 24 and week 48 (observation period) in patients who were successfully treated (observation period)
Variation of patient's global satisfaction using Likert score | 12 weeks
  Variation of patient's global satisfaction using Likert score at each follow-up visit
Variation of patient's global satisfaction using Likert score | 24 weeks
  Variation of patient's global satisfaction using Likert score at each follow-up visit
Variation of patient's global satisfaction using Likert score | 48 weeks
  Variation of patient's global satisfaction using Likert score at each follow-up visit
Variation of the physician global evaluation of treatment efficacy | 12 weeks
  Variation of the physician global evaluation of treatment efficacy on facial vitiligo using Likert score at each follow-up visit
Variation of the physician global evaluation of treatment efficacy | 24 weeks
  Variation of the physician global evaluation of treatment efficacy on facial vitiligo using Likert score at each follow-up visit.
Variation of the physician global evaluation of treatment efficacy | 48 weeks
  Variation of the physician global evaluation of treatment efficacy on facial vitiligo using Likert score at each follow-up visit.
Variation of the Dermatology Life Quality Index | 24 weeks
  Variation of the Dermatology Life Quality Index (DLQI) between inclusion and after 24 weeks of treatment between the 2 groups
Number of participants with Adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khaled EZZEDINE, Principal Investigator — University Hospital Bordeaux, France
Locations (4):
- France (4):
  - University Hospital of Bordeaux - St André Hospital, Bordeaux
  - Regional Hospital Center of Le Mans -, Le Mans
  - University Hospital Center of Nice - Hôpital de l'Archet, Nice
  - University Hospital Center of Rennes - Hôpital Pontchaillou, Rennes

REFERENCES:
- [Derived] Seneschal J, Duplaine A, Maillard H, Passeron T, Andreu N, Lassalle R, Favary C, Droitcourt C, Taieb A, Ezzedine K. Efficacy and Safety of Tacrolimus 0.1% for the Treatment of Facial Vitiligo: A Multicenter Randomized, Double-Blinded, Vehicle-Controlled Study. J Invest Dermatol. 2021 Jul;141(7):1728-1734. doi: 10.1016/j.jid.2020.12.028. Epub 2021 Feb 4. PMID 33549606